CLINICAL TRIAL: NCT06071455
Title: The Effect of Platelet-rich Fibrin and Vitamin Dꝫ Injections on Canine Retraction: A Randomized Controlled Clinical Trial
Brief Title: The Effect of Platelet-rich Fibrin and Vitamin Dꝫ Injections on Canine Retraction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Rehab Abd El Razek Abd El Aziz Khalil, lecturer of Orthodontics, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: # REC-FDBSU/06042023-03/AR
Record Dates: First submitted 2023-10-01; First posted 2023-10-06 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Acceleration of Tooth Movement
Keywords: Platelet-rich Fibrin; Vitamin D3; Canine retraction
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: split-mouth, prospective, single-center, single-blinded, two-arm randomized clinical trial with a 1:1 allocation ratio.
Who Masked: Outcomes Assessor
Masking Description: single-blinded limited to the outcome assessment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet-rich Fibrin (Experimental): A 20 ml blood sample will be drawn from the median cubital vein into a PRF tube. Centrifugation will be done at 700 rpm for 3 minutes and the liquid of PRF will be suctioned out using a separate syringe. PRF will be injected distal to the canine on the experimental side three times; at the beginning of canine retraction (T0), 1 month after the start of canine retraction (T1), and 2 months after the start of canine retraction (T2).
  Interventions: Other: Platelet-rich fibrin
- Vitamin D3 (Experimental): Subjects will receive vitamin Dꝫ injection distal to the canine on the experimental side three times; at the beginning of canine retraction (T0), 1 month after the start of canine retraction (T1), and 2 months after the start of canine retraction (T2).
  Interventions: Other: Vitamin D3

INTERVENTIONS:
Other: Platelet-rich fibrin — injected distal to the canine on the experimental side.
  Arms: Platelet-rich Fibrin
Other: Vitamin D3 — injected distal to the canine on the experimental side.
  Arms: Vitamin D3

SUMMARY:
the aim of this study is to assess and compare the effect of PRF and vitamin Dꝫ injection on the rate of canine retraction and to determine the bone thickness changes correlated with the two techniques.

DETAILED DESCRIPTION:
* Participants will be recruited from the Faculty of Dentistry, Beni-Suef University. All subjects will be informed of the treatment procedures and will sign a consent form.
* Subjects will be randomly divided into two groups:

Group 1 (PRF group): upper canine retraction will be facilitated by PRF injection that will be randomly assigned to one side (experimental side). The contralateral side will serve as the control one.

Group II (Vitamin Dꝫ group): canine retraction will be facilitated by Vitamin Dꝫ injection that will be randomly assigned to one side (experimental side). The contralateral side will serve as the control one.

* The predicted sample size (n) was a total of (28) cases (i.e. 14 cases per group). Sample size calculation was performed using G*Power version 3.1.9.7
* Randomization:

Simple randomization will be designed with the aid of a computer-generated schedule with 1:1 allocation ratio. Allocation concealment will be achieved using identical opaque, sealed envelopes. Randomization and allocation concealment will be performed by one of the academic staff who will not be involved in the study and will keep the allocation table away from the operators. The operator will shuffle the sealed envelopes and will ask the patient to pick one envelope at the time of recruitment. In each group, a randomly selected side will act as the experimental side while the contralateral side will serve as the control. Blinding of the operators will not be applicable and so blinding will be limited to the outcome assessment.

Methodology:

All patients will be treated with a 0.022-inch MBT bracket system. Leveling and alignment phase will be completed until a 0.017 X 0.025'' stainless steel wire will be inserted passively into the bracket slot. Before canine retraction, the subject will be randomly assigned to one of the groups (PRF or Vitamin Dꝫ group). In both groups, canine retraction will be performed with closed Ni-Ti coil springs with a force of 150 g per side that will be adjusted by the use of a force gauge.

PRF group:

A 20 ml blood sample will be drawn from the median cubital vein into a PRF tube. Centrifugation will be done at 700 rpm for 3 minutes and the liquid of PRF will be suctioned out using a separate syringe. PRF will be injected distal to the canine on the experimental side three times; at the beginning of canine retraction (T0), 1 month after the start of canine retraction (T1), and 2 months after the start of canine retraction (T2).

Vitamin Dꝫ group:

Subjects will receive vitamin Dꝫ injection distal to the canine on the experimental side three times; at the beginning of canine retraction (T0), 1 month after the start of canine retraction (T1), and 2 months after the start of canine retraction (T2).

* For both groups, alginate impressions will be taken just before canine retraction and at a monthly rate till the end of the canine retraction phase. Study casts will be obtained, and the rate of canine movement will be measured every month.
* Cone beam computed tomography (CBCT) will be obtained before treatment and after canine retraction to evaluate the bone thickness changes associated with the two techniques.
* The results will be obtained and statistically evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18- 40 years old.
2. Angle Class I or Class II dental malocclusion that required bilateral maxillary first premolar extraction and upper canine retraction as a part of the treatment plan.
3. Good to fair oral hygiene.
4. Normal probing depth.

Exclusion Criteria:

1. Active periodontal disease.
2. Poor oral hygiene.
3. Systemic diseases or medications that alter bone metabolism or tooth movement.
4. Craniofacial anomalies.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2023-05-11 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
evaluate the rate of upper canine retraction in the PRF (platelet-rich fibrin) and Vitamin Dꝫ groups and compare between them. | 3 - 4 months
  alginate impressions will be taken just before canine retraction and at a monthly rate till the end of the canine retraction phase. Study casts will be obtained, and the rate of canine movement will be measured every month.

SECONDARY OUTCOMES:
investigate the bone thickness changes associated with the two injection techniques and compare between them after canine retraction. | 6 months
  Cone beam computed tomography (CBCT) will be obtained before treatment and after canine retraction to evaluate the bone thickness changes associated with the two techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Rehab Khalil, Principal Investigator — Faculty of Dentistry, Beni Suef University
Locations (1):
- Faculty of Dentistry Beni Suef University, Banī Suwayf, Beni Suef Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta P, Bhagyalakshmi A, Avinash BS, Prashant A, Raghunath N. Evaluation of injectable platelet-rich fibrin effect on the rate of canine retraction and alkaline phosphatase levels: An in-vivo study. Am J Orthod Dentofacial Orthop. 2022 Nov;162(5):735-743. doi: 10.1016/j.ajodo.2021.07.019. Epub 2022 Aug 23. PMID 36008239
- [Background] Erdur EA, Karakasli K, Oncu E, Ozturk B, Hakki S. Effect of injectable platelet-rich fibrin (i-PRF) on the rate of tooth movement. Angle Orthod. 2021 May 1;91(3):285-292. doi: 10.2319/060320-508.1. PMID 33459765
- [Background] Cagli Karci I, Baka ZM. Assessment of the effects of local platelet-rich fibrin injection and piezocision on orthodontic tooth movement during canine distalization. Am J Orthod Dentofacial Orthop. 2021 Jul;160(1):29-40. doi: 10.1016/j.ajodo.2020.03.029. Epub 2021 May 4. PMID 33962809
- [Background] Zeitounlouian TS, Zeno KG, Brad BA, Haddad RA. Effect of injectable platelet-rich fibrin (i-PRF) in accelerating orthodontic tooth movement : A randomized split-mouth-controlled trial. J Orofac Orthop. 2021 Jul;82(4):268-277. doi: 10.1007/s00056-020-00275-x. Epub 2021 Jan 22. PMID 33481053
- [Background] Reyes Pacheco AA, Collins JR, Contreras N, Lantigua A, Pithon MM, Tanaka OM. Distalization rate of maxillary canines in an alveolus filled with leukocyte-platelet-rich fibrin in adults: A randomized controlled clinical split-mouth trial. Am J Orthod Dentofacial Orthop. 2020 Aug;158(2):182-191. doi: 10.1016/j.ajodo.2020.03.020. Epub 2020 Jun 24. PMID 32591274
- [Background] Varughese ST, Shamanna PU, Goyal N, Thomas BS, Lakshmanan L, Pulikkottil VJ, Ahmed MG. Effect of Vitamin D on Canine Distalization and Alveolar Bone Density Using Multi-slice Spiral CT: A Randomized Controlled Trial. J Contemp Dent Pract. 2019 Dec 1;20(12):1430-1435. PMID 32381845
- [Background] Al-Attar A, Abid M. The Effect of Vitamin D3 on the Alignment of Mandibular Anterior Teeth: A Randomized Controlled Clinical Trial. Int J Dent. 2022 Feb 14;2022:6555883. doi: 10.1155/2022/6555883. eCollection 2022. PMID 35198025
- [Background] Khalaf RM, Almudhi AA. Effects of vitamin D deficiency on the rate of orthodontic tooth movement: An animal study. Saudi Dent J. 2022 Feb;34(2):129-135. doi: 10.1016/j.sdentj.2021.12.008. Epub 2021 Dec 23. PMID 35241902